CLINICAL TRIAL: NCT02447601
Title: An Open-label,Sequential,Single-site Study to Evaluate the Pharmacokinetics of Simvastatin When Coadministered With Polyethylene Glycol Loxenatide (PEX168) in Healthy Adult Subjects
Brief Title: Evaluate the Pharmacokinetics of Simvastatin When Coadministered With PEX168 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PEX168-Ik; PEX168-Ik (Other: JiangsuHaosen)
Record Dates: First submitted 2015-03-25; First posted 2015-05-19 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — polyethylene glycol loxenatide; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Simvastatin and PEX168(200µg) (Experimental): Simvastatin: 40mg, oral Administration. PEX 168: 200µg,injected subcutaneously,once a week.
  Interventions: Drug: PEX168; Drug: Simvastatin

INTERVENTIONS:
Drug: PEX168 — 200µg,injected subcutaneously,once a week.
  Other Names: Polyethylene Glycol Loxenatide
Drug: Simvastatin — 40mg,oral,two times
  Other Names: Shujiangzhi

SUMMARY:
To assess the effect of PEX168 doses on the pharmacokinetics of simvastatin(as determined by simvastation acid) in healthy subjects.

To assess the safety of single doses of simvastation administered with and without PEX168

DETAILED DESCRIPTION:
This was an open-label, sequential, single-center study that evaluated the pharmacokinetics of simvastatin when coadministered with PEX168 in healthy adult subjects. The total duration of each subject's participation in the study was approximately 10 weeks, which included up to a 14-day Screening Period, a 34-day Treatment Period, and an approximately 4-week Follow-up Period.

Center: This study was conducted at a single site in Shanghai Mental Health Center (SMHC)of China Treatment.All subjects receives a single 40-mg oral dose of simvastatin on Day 1 followed by 5 weekly 200μg doses of PEX168 injected subcutaneously beginning on Day 3 and a second single 40-mg oral dose of simvastatin on Day 33.

ELIGIBILITY:
Inclusion Criteria:

An individual who met all of the following criteria was eligible for the study.

1. Healthy male aged 18 to 45 years (including both ends) at the time of signing the informed consent.
2. Weighing not less than 50kg，Body Mass Index (BMI)of 18 to 25kg/m2.
3. No history of cardiovascular, liver, kidney, gastrointestinal, neuropsychiatric and other diseases, no history of drug allergy.
4. Capable of giving written informed consent, which included compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. Known for any study drug allergy (PEX168, simvastatin) or similar drug allergy (GLP-1 receptor agonists, GLP-1 analogue, statins) or allergic constitution;
2. Having Alcohol and drug abuse within first 6 months before screening;
3. Smoked within 3 months before screening;
4. Received GLP-1 receptor agonists, GLP-1 analogs, DPP-IV inhibitors, or any other similar structure drug for treatment before screening;
5. Following a thorough medical examination, clinically significant abnormalities were found;
6. In screening period, blood pressure greater than 140 / 90mmHg, retest after diagnosis or pulse rate is higher than 100bpm person;
7. In screening period, ECG QTc> 450ms, diagnosed after retest;
8. In screening period, serum creatinine or urine protein is abnormal, and were determined to be clinically significant by the investigator;
9. In screening period, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), γ- glutamate GGT (γ-GT), total bilirubin (Tbil) is greater than the normal range limit, and investigator determines to have clinical significance;
10. In screening period, creatine kinase (CK) exceeds the upper limit of the normal range, and judged by the investigator to be clinical significant;
11. In screening period, having thyroid dysfunction;
12. Before screening there is a history of medullary thyroid cancer;
13. Having any surgery (including the impact of gastric emptying of gastrointestinal surgery) within 6 months before screening;
14. Participate in blood donation and donation amount ≥400ml within three months before screening, or who participate in blood donation or blood transfusion within a month;
15. Using any of the tested drugs may affect prescription drugs, nonprescription drugs, herbs, food (such as grapefruit juice) or food supplements persons 2 weeks before screening;
16. Drinking medication or caffeine-containing xanthine food and beverage (listed in annex 3), strenuous exercise, or other effects of drug absorption, distribution, metabolism, excretion and other factors 2 days before screening.
17. Any clinically significant by the investigator determined that acute diseases before Screening occurred within a month too;
18. There is a history of pancreatitis or acute pancreatitis before screening;
19. Having dyslipidemia, coronary heart disease, and a history of high cholesterol before screening.
20. There are lung disease histories, history of chronic liver and gallbladder disease, cholecystitis history, history of bladder disease, a history of colon inflammation before screening.
21. Within three months before screening participated in any drug or medical device clinical trials were (including placebo);
22. Hepatitis B surface antigen, hepatitis C antibody, HIV antibody, syphilis antibody test positive;
23. Reluctant to take effective contraceptive methods of contraception. During the trial, there was family planning within six months after their spouses during the trial or the last dose (first 33 days);
24. The investigator believe that any situation that might lead to any subject cannot be completed or to the subject of this study bring significant risk.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2015-05-14 (Actual); Study Completion 2015-08-11 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of simvastatin and simvastatin acid. | Baseline to Day34
  Plasma concentrations of simvastatin and simvastatin acid, and to calculate the pharmacokinetic parameters: Tmax, Cmax, AUC0-t, AUC0-∞, λz, t1 / 2, Vd / F, CL / F, etc.

SECONDARY OUTCOMES:
Incidence of adverse events and serious adverse events | Baseline to Day67

CONTACTS AND LOCATIONS:
Overall Officials: Huafang Li, MD, Principal Investigator — Shanghai Mental Health Center (SMHC)
Locations (1):
- Shanghai Mental Health Center (SMHC), Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No